CLINICAL TRIAL: NCT03176030
Title: Can Fortified Foods Improve Energy and Protein Intake in Older People Whilst in Hospital? A Pilot Study
Brief Title: Fortified Foods in Older Inpatients
Status: Withdrawn | Type: Observational
Why Stopped: Study team submitted IRAS form and the ethic committee advised that this pilot study is more service evaluation and no REC ethical approval was required.
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: RHM MED1428
Record Dates: First submitted 2017-05-16; First posted 2017-06-05 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Malnutrition; Dementia; Aging; Frail Elderly Syndrome
MeSH Terms: conditions — Malnutrition; Dementia | interventions — Food, Fortified

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fortified foods: Fortified foods will be delivered to this group for 3 consecutive days mainly on a mid-meal trolley three times a day (between breakfast and lunch around 10am, between lunch and dinner around 3 pm, and in the evening). However, fortified foods will be available 24 hours and patients will be encouraged to order as many as they like anytime during the day.
  Interventions: Dietary Supplement: Fortified Foods
- Baseline: Prior to implementing the intervention, dietary intake among eligible patients offered the standard hospital menu will be measured on the study wards for 24 hours during three days in each of the study wards to estimate the energy and protein intake.

INTERVENTIONS:
Dietary Supplement: Fortified Foods — The intervention under study is the provision of between-meal fortified foods (enhanced with protein, energy, and micronutrients) and meal supplementation where meals are poorly consumed. Foods will include both savory and sweet foods with different flavors. Foods will be matched as closely as possible in protein and energy and are calculated to provide typically 210 kcal and 5g protein per item. The volume / weight of the foods are standardized to be of relatively small portion size, such as 100 ml for ice-creams, 40 g for cakes and biscuits, and 100 ml for soup. Some of the products will be supplemented with micronutrients particularly needed by older adults, such as Vitamins (C, D, folic acid, B2, B6) and calcium at one third of the Dietary Reference Values (DRV) per portion. The aim is to achieve a daily consumption of two additional fortified food items.
  Groups: Fortified foods

SUMMARY:
Malnutrition in older inpatients is a significant problem espicially among those with dementia. A number of methods have been used to tackle this issue and oral nutritional supplements (ONS) were proven to be the most effective way. However, they are limited by their poor tolerability due to lack of familiarity with these products. An alternative method is to fortify familiar food with protein, energy and micronutrient. thus, the aim of this study to test the feasibility and acceptability of delivering fortified foods to older patients whilst in hospital including those with dementia and frailty. This pilot study will compare the daily protein and energy intake in older people before and after offering fortified food. Furthermore, patients' likeability and staff acceptability of these fortified foods will be assessed.

DETAILED DESCRIPTION:
Malnutrition is a significant problem amongst hospitalised older people, and can impede effective recovery. Oral nutritional supplements (ONS) are limited by their poor tolerability and an alternative strategy is food fortification, the addition of protein/energy/micronutrients to frequently eaten food. The aim of this pilot study is to establish the feasibility and acceptability of delivering fortified foods to older people including those who have dementia and frailty whilst in hospital and to assess whether fortified foods could increase the energy and protein intake.

This is a quasi-experimental study on acute medical wards for older inpatient in two UK hospitals, with a before and after comparison. The intervention involves the provision of additional between-meal fortified foods (enhanced with protein, energy, and micronutrients) and meal supplementation. Daily energy and protein intake will be assessed for three consecutive days during the baseline period and then in the intervention period. Likeability of fortified food and food choices (the number, type, and frequency of fortified foods consumed) will be examined. Likeability of fortified food by patients will be assessed using likeability scales. Interviews or focus groups will be conducted with staff to assess the acceptability of fortified food. Costs related to developing, packing and delivering the fortified foods will be calculated.

The findings of this pilot study will identify whether delivering fortified food is feasible in acute elderly care wards, which foods are preferred and their acceptability. The results will inform the design of a definitive clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Both female and male participants in each hospital.
2. Patients aged 70 years and above including those who have dementia and frailty.

Exclusion Criteria:

1. Patients receiving enteral tube feeding or parenteral nutrition
2. Patients with a known food allergy, eating disorder or illness, which requires a therapeutic diet incompatible with fortification.
3. Patients who are receiving end of life care.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Eligible patients will be female and male older patients who are admitted to acute medical wards for older people in two hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Daily energy and protein intake | 3 consecutive months
  Daily dietary intake will be assessed on three days during both the baseline and intervention periods using visual assessment. each food or meal will be weighed before serving and once the patient has finished using calibrated scales. In addition, a photograph of each plate of food will be taken before and after consumption for each eligible patient. At the end of each meal, the proportion of uneaten (leftover) food will be recorded in quartiles (0%, 25%, 50%, 75%, or 100%) for each component
Feasibility of delivering fortified foods | 3 days intervention period
  The number, type, and frequency of fortified foods chosen by eligible patients during the intervention period will be recorded. This will be done by using a food chart with images. Thus data will be collected on the type of foods (ice-creams, biscuits, soups or cakes) chosen, flavors preferred by individual patients initially and repeat choices, the number of foods chosen each time and at which time of the day.
Patient's likeability of fortified foods | 3 days intervention period
  A 9-point likeability scale will be completed for each eligible patient to test likeability of fortified foods after each meal or snack time during the intervention period.

SECONDARY OUTCOMES:
Acceptability of fortified food | within 4 weeks of completing the intervention
  A purposive sample staff (nursing staff, catering staff and volunteers) involved in the delivery of fortified foods from the study wards in both hospitals will be invited to take part in interviews or focus groups. Participants will be recruited until theoretical saturation has been met; a total sample of approximately 15-20 staff members across the two settings is anticipated to be adequate.

CONTACTS AND LOCATIONS:
Locations (1):
- Southampton Genral Hospital, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data will be shared unless requested directly from authors